CLINICAL TRIAL: NCT05880966
Title: Functional Training for Overweight/obese Adults with Mobility-related Disabilities
Brief Title: Functional Fitness for Overweight or Obese Adults with Mobility Disabilities
Acronym: COBRE Pilot
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Kansas (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 00043722
Record Dates: First submitted 2023-04-17; First posted 2023-05-30 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2024-06

CONDITIONS: Mobility Limitation; Overweight or Obesity; Physical Disability
MeSH Terms: conditions — Mobility Limitation; Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- COBRE Single Group (Experimental): All participants will complete the 6-mos functional fitness interventions
  Interventions: Behavioral: Functional Fitness

INTERVENTIONS:
Behavioral: Functional Fitness — Six month, thrice weekly functional fitness sessions will include a warm-up (15 minutes), skill or strength work (30 minutes) and a cool down (15 minutes)

SUMMARY:
Over 64 million people in the U.S. have a permanent disability, with mobility-related disability (MRD) representing the most prevalent disability type (13.7%). Adults with MRD are 66% more likely to be overweight or obese than their non-disabled peers. Exercise in adults with MRD is important for weight management and is associated with improvements in obesity-related health conditions including hypertension, hyperlipidemia, insulin processing/sensitivity, etc. However, over half (57%) of adults with MRD do not exercise, while 22% engage in exercise of insufficient duration or intensity to obtain health benefits. Adults with MRD face numerous barriers to participation in community-based exercise, and exercise is frequently limited to short-term referrals for outpatient physical and/or occupational therapy. High-intensity functional training (HIFT) represents a potentially effective strategy for community-based exercise to support body weight and obesity-related health conditions, in addition to improving physical function and aspects of psychosocial health for people with disabilities. Preliminary evidence supports the effectiveness of HIFT to improve body composition, cardiovascular and muscular fitness, insulin processing and insulin sensitivity in non-disabled adults who are overweight/obese. To date, no study has systematically evaluated the feasibility or effectiveness of a community-based HIFT intervention for improving obesity-related health outcomes in overweight/obese adults with MRD. Thus, the proposed study will implement a 6-mo. pilot trial to evaluate the feasibility and potential effectiveness of a HIFT intervention (60 min sessions/3 days/wk.) in 25 adults with MRD and overweight/obesity.

This study will address the following aims:

Aim 1: Evaluate the intervention feasibility based on participant recruitment, session attendance, retention, outcome assessment completion, and the results of semi-structured exit interviews to obtain information regarding experience and overall satisfaction with the intervention.

Aim 2: Evaluate changes (baseline - 6 mos.) in weight and fat-mass/fat-free mass, and components of the metabolic syndrome (waist circumference, blood pressure, HDL-cholesterol, triglycerides, fasting glucose).

DETAILED DESCRIPTION:
Over 64 million people in the U.S. have a permanent disability, with mobility-related disability (MRD) representing the most prevalent disability type (13.7%). The occurrence of chronic conditions including obesity, diabetes, hypertension, and hyperlipidemia are significantly higher in adults with disabilities compared with non-disabled adults. Adults with MRD are 66% more likely to be overweight or obese than their non-disabled peers. Exercise in adults with MRD is important for weight management and is associated with improvements in obesity-related health conditions including hypertension, hyperlipidemia, insulin processing/sensitivity, etc. However, over half (57%) of adults with MRD do not exercise, while 22% engage in exercise of insufficient duration or intensity to obtain health benefits. Adults with MRD face numerous intrapersonal, environmental, and financial barriers to participation in community-based exercise, and exercise is frequently limited to short-term referrals for outpatient physical and/or occupational therapy. While effective, these clinical settings do not provide a long-term strategy for the delivery of exercise programs to the general population of adults with MRD.

High-intensity functional training (HIFT) represents a potentially effective strategy for community-based exercise to support body weight and obesity-related health conditions, in addition to improving physical function and aspects of psychosocial health for people with disabilities. HIFT incorporates multiple exercise modalities and constantly varied functional movement patterns designed to simulate daily activities (e.g., sit-to-stand, transferring). The variety of functional movements offered by HIFT may be more enjoyable and result in better long-term adherence compared with traditional single mode continuous aerobic exercise such as stationary biking, arm cycling, or treadmill walking/running. Preliminary evidence supports the effectiveness of HIFT to improve body composition, cardiovascular and muscular fitness, insulin processing and insulin sensitivity in non-disabled adults who are overweight/obese. The limited available data relative to HIFT interventions in adults with MRD provides some support for the feasibility and potential effectiveness of HIFT in adults with MRD including high retention rates, positive intervention experiences, improved functional capacity and confidence in performing daily movements. However, this data is based on unpowered pilot studies and unpublished these/dissertations with poor descriptions of the HIFT interventions, and thus should be cautiously interpreted. To date, no study has systematically evaluated the feasibility or effectiveness of a community-based HIFT intervention for improving obesity-related health outcomes in overweight/obese adults with MRD. Thus, Thus, the proposed study will implement a 6-mo. pilot trial to evaluate the feasibility and potential effectiveness of a HIFT intervention (60 min sessions/3 days/wk.) in 25 adults with MRD and overweight/obesity. The intervention will be conducted at two community-based facilities in greater Kansas City that have been conducting HIFT sessions for adults with disabilities for over three years. HIFT sessions will be delivered by instructors certified by the Adaptive Training Academy (ATA), a non-profit organization, which provides training in adapting and conducting safe HIFT sessions for people with disabilities. This study will address the following aims:

Aim 1: Evaluate the intervention feasibility based on participant recruitment, session attendance, retention, outcome assessment completion, and the results of semi-structured exit interviews to obtain information regarding study improvements, perceptions of the length/frequency of the intervention, satisfaction with instructors, exercise facilities, session content, difficulties with compliance, and overall satisfaction with the intervention.

Aim 2: Evaluate changes (baseline - 6 mos.) in weight (primary outcome), and secondary outcomes including fat-mass/fat-free mass, and components of the metabolic syndrome (waist circumference, blood pressure, HDL-cholesterol, triglycerides, fasting glucose). Energy expenditure will also be measured during HIFT sessions using portable indirect calorimetry.

Results from this study will inform the development of an NIH-R01 application to conduct an adequately powered, randomized trial in overweight/obese adults with MRD to evaluate the effectiveness of HIFT over a longer time frame (i.e., 12 mos.), on the obesity-related outcomes proposed for this study plus additional health and functional related outcomes. If ultimately shown to be effective, the physical infrastructure available in the over 5,000 HIFT affiliates across the country would provide the framework for widespread adoption, implementation, and maintenance of inclusive HIFT programs for adults with MRD.

ELIGIBILITY:
Inclusion Criteria:

* 18-64 years of age
* Have a permanent disability that affects mobility (1 year +);
* Body mass index between 24-52
* Never been a part of a functional fitness program before
* Have no significant health impairment that would contraindicate exercise (physician clearance required)
* Serve as their own guardian

Exclusion Criteria:

* Younger than 18 years of age or 65 years or older
* Have a disability that was acquired within 1 year of starting the study or has a non-permanent mobility limitation (e.g., broken arm);
* Have a body mass index less than 24 or greater than 52
* Has previously been involved in functional fitness
* Unable to obtain physician clearance
* Are not their own guardian

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-04-17 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Weight | Change from Baseline weight at 6 months (post-intervention)
  Weight will be measured in duplicate using a portable calibrated, digital scale to the nearest 0.1 kg.

SECONDARY OUTCOMES:
Body Composition | Change from Baseline body comp at 6 months (post-intervention)
  Fat free and fat-mass Dual Energy X-ray Absorptiometry (DEXA) will be performed at the KU Edwards campus to determine the fat-free mass, fat mass, and body fat percentage (Prodigy Advance Plus, GE, Madison, WI)
Waist Circumference | Change from Baseline waist circumference at 6 months (post-intervention)
  Waist circumference will be assessed with a calibrated tape. For those unable to stand, waist circumference will be measured in the seated position at the umbilicus. Three measurements will be obtained with the outcome recorded as the average of the closest 2 measures.
Blood Pressure | Change from Baseline blood pressure (diastolic and systolic) at 6 months (post-intervention)
  Blood pressure will be obtained with an automated sphygmomanometer (DinaMap ProCare 100, General Electric) using the NHANES blood pressure protocol and recommendations of the American Heart Association.
Glucose | Change from Baseline fasting glucose at 6 months (post-intervention)
  Fasting glucose will be assessed following finger prick blood draw with 8 hours prior of fasting
Cholesterol | Change from Baseline HDL cholesterol at 6 months (post-intervention)
  HDL Cholestserol will be assessed following finger prick blood draw
Triglycerides | Change from Baseline triglycerides at 6 months (post-intervention)
  Triglycerides will be assessed following finger prick blood draw
Body Mass Index | Change from Baseline BMI at 6 months (post-intervention)
  Weight will be measured in duplicate using a portable calibrated, digital scale to the nearest 0.1 kg. Height will be measured in meters, and body mass index (BMI) will be calculated with the following formula: kg/m2
Perceived Quality of Life | Change from Baseline QOL at 6 months (post-intervention)
  World Health Organization Quality of Life an internationally recognized and established short measure assessing quality of life. There are 26 items on this survey, with a minimum value of 26, and a maximum value of 130. The higher the score, the higher the perceived quality of life.
Perceived Life Satisfaction | Change from Baseline life satisfaction at 6 months (post-intervention)
  the Satisfaction with Life Questionnaire will be used as an additional assessment of well-being. There are five items on this survey, with a minimum score of 5 and a maximum score of 35, higher scores indicate higher satisfaction with life.
Flexibility | Change from Baseline flexibility at 6 months (post-intervention)
  Back Scratch Test - 1 arm above the head, bent elbow, reach down across the back as far as possible. Simultaneously, the opposite arm bent at elbow and forearm is extended up along the back as far as possible to that the fingers of both hands meet or overlap. The distance of overlap or the distance between the tips of the middle fingers is measured in centimeters.
Balance (Seated) | Change from baseline balance at 6 months (post-intervention)
  Participants who are non-ambulatory participants will complete the Function in Sitting Test. Minimum score is 0 and maximum score is 56, where higher scores indicate better balance.
Balance (standing) | Change from baseline balance at 6 months (post-intervention)
  Participants who are ambulatory will complete the Berg Balance Scale test. Minimum score is 0 and maximum score is 56, where higher scores indicate better balance.
Strength | Change from baseline strength at 6 months (post-intervention)
  Grip Strength with dynameter. Participants will be seated with elbow flexed at 90 degrees, forearm in a neutral position and write between 0 and 30 degrees of flexion. participants will use their dominant hand and the 5 second squeeze will occur in duplicate, with 15 second rest in between and the score averaged to the nearest 0.1 kg.
Mobility | Change from baseline mobility at 6 months (post-intervention)
  participants who are ambulatory will complete the 6-minute walking test and the 10-meter walking speed test, both of which can be completed with the help of an assistive device as needed. Distance covered during the 6-minute walking test will be calculated with meters, and average walking speed will be calculated as miles per hour. Participants who are non-ambulatory will complete a 6-minute push test and the Timed Forward Wheeling (23-meters) test. Distance covered during the 6-minute push test will be converted to meters, and timed forward wheeling will assess average speed calculated as miles per hour.
Sense of Community | Change from baseline sense of community at 6 months (post-intervention)
  The Sense of Community Scale will be used to assess perceptions of community among the administration, social spaces, other members and competition. Minimum score is 18 and maximum score is 72, where higher scores indicate greater sense of community.
Shoulder Pain - manual wheelchair users only | Change from baseline shoulder pain at 6 months (post-intervention)
  he Wheelchair User's Shoulder Pain Index will be used to assess self-report changes in shoulder pain during daily functional activities with a 10-point visual analog scale. Minimum score is 15 and maximum score is 150, where higher scores indicate greater pain.
Exercise self-efficacy | Change from baseline self-efficacy at 6 months (post-intervention)
  28-item Self-Related Abilities for Health Practices Scale to assess self-efficacy scores regarding exercise, nutrition, health practices and psychological well-being. Minimum score is 0 and maximum score is 112, where higher scores indicate greater exercise self-efficacy.
Sleep | Change from baseline sleep at 6 months (post-intervention)
  Sleep Disturbance Short Form (PROMIS Health Organization, 8b) will be used to assess self-report sleep quality in the past 7 days. Minimum score is 8 and maximum score is 40, where lower scores indicate better sleep.
Barriers to Health | Change from baseline perceived barriers at 6 months (post-intervention)
  The 16-item Barriers to Health Adapted for People with Disabilities will assess participant self-report of perceived motivational and external barrier to exercise. Minimum score is 18 and maximum score is 72, where higher scores indicate greater perceived barriers to health promoting activities.
Psychological Need Satisfaction | Change from baseline perceived need satisfaction at 6 months (post-intervention)
  The Psychological Need Satisfaction in Exercise Questionnaire will be used to assess need satisfaction within the functional fitness environment. Include three subscale autonomy, competence, and relatedness. Minimum score is 18 and maximum score is 108, where higher scores indicate better need satisfaction.
Self-determination | Change from baseline perceived need self-determination at 6 months (post-intervention)
  Behavioral Regulation in Exercise Questionnaire will assess changes to perceived behavioral regulation (autonomous vs. external regulation) with in the functional fitness environment. 19 items with 5 subscales (external, introjected, identified, and intrinsic). Minimum score is 19 and maximum score is 95, where higher scores indicate more self-determined motives for exercise.
Perceived Functional Performance | Change from baseline perceived performance in occupational activities at 6 months (post-intervention)
  The Canadian Occupational Therapy Measure is a valid and reliable standardized assessment used to identify occupational performance problems experienced by a client. Performance areas report by the client as challenging or unable to do will be documented in a list. Then the client will rate the perceived importance of each problem area on the list. Only the most important performance areas (top five maximum) will be included in the COPM assessment. The client will then rate their current performance ability for each of these performance areas. The client's ratings of performance ability will be used to calculate the client's baseline average occupational performance ability. Baseline average performance scores are then used to determine if a client's occupational performance improvements occur over time. Range of scoring is 1-10, where higher scores indicate greater perceived performance.
Perceived Functional Performance | Change from baseline perceived satisfaction in performing occupational activities at 6 months (post-intervention)
  The Canadian Occupational Therapy Measure is a valid and reliable standardized assessment used to identify occupational performance problems experienced by a client. Performance areas report by the client as challenging or unable to do will be documented in a list. Then the client will rate the perceived importance of each problem area on the list. Only the most important performance areas (top five maximum) will be included in the COPM assessment. The client will then rate their current satisfaction of their ability for each of these performance areas. The client's ratings satisfaction will be used to calculate the client's baseline average occupational satisfaction of their ability. Baseline average satisfaction scores are then used to determine if a client's occupational performance improvements occur over time. Range of scoring is 1-10, where higher scores indicate greater perceived satisfaction.

OTHER OUTCOMES:
Energy expenditure | Week 12 of the intervention - one time exploratory measure
  energy expenditure will be assessed at two, randomly selected sessions for each participant. This will be done using a previously validated portable, open-circuit indirect calorimeter (Cosmed, Italy) which measures breath-by-breath ventilation, expired oxygen, and carbon dioxide. The flow turbine will be calibrated using a 3.0-L syringe. The lightweight (~1.5 kg) portable system will be attached by a harness around the waist and shoulders of the participant before each assessment. During exercise sessions, participants will breathe into a facemask that directs air into the unit housing the O2 and CO2 analyzers. Data will be retrieved for analysis via a serial port interface and software provided with the calorimeter and aggregated over 20-second epochs for the calculation of 1-min averages.
Attendance | Observed each week of the 24-week intervention
  Participant attendance for the functional fitness sessions will be recorded
Work Capacity | Change in baseline work capacity (time; A1) at 12 weeks and 24 weeks of the intervention
  Participants will complete work capacity testing during week 2, 12, and again at week 24. Work capacity (A1) will be assessed by the outcome measure of time to complete the benchmark exercise session - in minutes and seconds. Lower times indicate improved work capacity.
Work Capacity | Change in baseline work capacity (reps; A2) at 12 weeks and 24 weeks of the intervention
  Participants will complete work capacity testing during week 2, 12, and again at week 24. Work capacity (A2) will be assessed by number of rounds and repetitions completed during the exercise session in a given amount of time. Higher rounds and repetitions indicate improved work capacity.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Kansas, Lawrence, Kansas, United States

IPD SHARING:
Plan to Share IPD: No